CLINICAL TRIAL: NCT01766180
Title: Association Between Fruitflow-II Treatment (Alone or in Combination With Resveratrol) and Changes in Cerebral Blood Flow, Fitness and Cognitive Function in Adults With Memory Complaints
Brief Title: Cerebrovascular and Cognitive Improvement by Resveratrol (resVida) and Fruitflow-II (CCIRF-II)
Acronym: CCIRF-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurolgy Institute for Brain Health and Fitness (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Majid Fotuhi, MD, PhD, Founder and Medical Chief Officer, Neurolgy Institute for Brain Health and Fitness
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-1048
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Memory Impairment
Keywords: Memory; Fruitflow; Resveratrol (resVida); Cerebral blood flow; Cardiopulmonary exercise test; Maximal VO2
MeSH Terms: conditions — Memory Disorders | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo / Placebo (No Intervention): In this control group, subjects receives placebo supplement pills without Fruitflow or ResVida ingredients.
- Fruitflow-II / Placebo (Active Comparator): In this group subjects receive Fruitflow-II daily supplied in capsules which contain 150 mg active ingredient. They also receive placebo capsules for resVida.
  Interventions: Drug: Fruitflow-II
- Placebo / resVida (Active Comparator): In this group subjects receive resVida daily supplied in capsules which contain 150 mg active ingredient. They also receive placebo capsules for Fruitflow-II.
  Interventions: Drug: resVida
- Fruitflow-II / resVida (Active Comparator): In this group subjects receive resVida and Fruitflow-II daily supplied in capsules which contain 150 mg active ingredient.
  Interventions: Drug: Fruitflow-II; Drug: resVida

INTERVENTIONS:
Drug: Fruitflow-II — 150 mg/day for 3 months, orally
  Arms: Fruitflow-II / Placebo; Fruitflow-II / resVida
Drug: resVida — 150 mg/day for 3 months, orally
  Other Names: "resVida" is other name for Resveratrol.
  Arms: Fruitflow-II / resVida; Placebo / resVida

SUMMARY:
The purpose of this study is to determine whether Fruitflow-II, Resveratrol (resVida), alone or in combination, are effective in the treatment of memory problems in adult patients with memory impairment. We also evaluate effects of these medications on blood flow to the brain and fitness, to find whether the possible improvement in memory is associated with the alterations in these parameters.

DETAILED DESCRIPTION:
Accumulating evidence suggests that tomato consumption has cardiovascular benefits, primarily through increasing blood flow in vivo; the active ingredient in tomato, or its extract (Fruitflow) have been shown to inhibit glycoprotein IIb/IIIa, similar to aspirin (which has antiplatelet activity and is used for secondary prevention of cardiovascular and cerebrovascular events in patients). Considering the fact that Fruitflow can improve the platelet function and peripheral blood flow, we hypothesized that Fruitflow can also increase the blood flow in the brain and thereby possibly enhance memory and cognitive function in middle-aged or elderly people who have memory complaints. Therefore, the initial goal of our study is to evaluate the effects of Fruitflow on brain blood and cardiovascular function by using Transcranial Doppler ultrasound (to check for changes in cerebral blood flow), cardiovascular fitness testing (to check for changes in VO2-max and stroke volume), and neurocognitive evaluation (to check for changes in memory and executive function).

Many pathways such as inflammation and oxidative stress are involved in the pathophysiology of memory loss with ageing. Recent studies have shown that a natural compound found in the skin of red grapes and also in wine, called "Resveratrol", have beneficial effects for prevention of cognitive decline by reducing inflammation and improving cardiovascular function. Therefore, our next goal is to evaluate whether administration of Resveratrol, by itself or in combination with Fruitflow, can improve brain blood flow, VO2-max, and cognitive performance.

Thus our clinical trial will have the following 4 arms: Fruitflow, Resveratrol, Fruitflow/Resveratrol combination, and placebo for each supplement.

The results of the study will potentially provide evidence that these natural supplements can have significant cardioprotective and neuroprotective properties in middle-aged and elderly adults.

Subjects (between 50 and 80 years old) complaining of memory problem who have MMSE (Mini-Mental State Examination) above 27 will be recruited from patients of Dr. Majid Fotuhi (PI at the Neurology Institute for Brain Health and Fitness). Flyers at the institute and advertisement in Baltimore will provide information about the opportunity to enroll in an observational study for 3 months, along with eligibility criteria. Participants will continue to receive routine and standard care, while data on outcome (i.e., dependent) variables and mediators will be collected over three study visits:

Day 1: at the onset of their participation: Assessment of memory and Cardiovascular Fitness Testing (CFT)

Day 2: Blood Test and Transcranial Doppler (TCD) Ultrasound at time 0 and 3 hours after taking the first dose of the supplements;

Month 3: Assessment of memory, Cardiovascular Fitness Testing, and Transcranial Doppler Ultrasound 3 months after daily treatment with supplements in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 50 and 80;
2. Having a primary care physician;
3. Ability to speak, read, and write English;
4. Logical Memory subtest (of the Wechsler Memory Scale - IV [WMS-IV]) raw score one standard deviation or greater below the mean of a younger population;
5. Be in stable overall health based on medical history and physical examination;
6. Sedentary or moderately active (< 2 aerobic session / week);
7. Suspend, for at least one month before participating in the study, the use of dietary supplements (fish oil, seed oils, ginkgo biloba, ginseng, resveratrol, fruit powder extracts and DHA; subjects who have high intake of these products are asked to take off these products for 4 weeks and after this washout period they will be recruited in the study). No more than one multivitamins per day is acceptable;
8. Wine intake not more than 2 glasses per day

Exclusion Criteria:

1. Patients reporting severe depression with or without suicidal ideation [Beck Depression Inventory (BDI) > 30 and BDI item #9 >1];
2. Patients with a severe language or hearing and/or vision impairment;
3. Pregnancy;
4. Patients presenting with delirium, dementia, or cognitive impairment (Mini-Mental Status Examination score < 26);
5. Current alcohol or substance abuse/dependence;
6. Major neurological and psychiatric diseases including Parkinson's disease, Alzheimer's disease, epilepsy, multiple sclerosis, concussion/traumatic brain injury, schizophrenia, bipolar disorder, psychosis, eating disorders;
7. Uncontrolled high blood pressure (> 180/100 mmHg) or a documented record of uncontrolled high blood pressure-related complications such as cerebral vascular disease (CVD), and/or large strokes with disability, uncontrolled diabetes mellitus (medical report of blood HbA1c > 7 during the last three months; in diabetic patients without this record HbA1c will be measured in the first blood testing), or history of major cardiopulmonary disease such as congestive heart failure, pulmonary disorders (COPD [emphysema or chronic bronchitis] and pulmonary embolism);
8. Documented evidence of the following findings in the current medical history of subjects:

   8-1- Low platelet number (< 170 x 10^9/ L); 8-2- Hematocrit below 40% for males or 30% for females; 8-3- Haemoglobin below 120 g/L for males or 110 g/L for females; 8-4- Prothrombin time (PT) values outside normal range of approximately 10-16 s;
9. Current hepatic failure, renal failure, bleeding disorders (hemophilia, Von Willebrand disease, esophageal varicoses);
10. Subjects who have given 500 ml of blood or more for transfusion purposes in the past month before entry into the study
11. Patients who take aspirin more than 325 mg/day
12. Current medications for cognition such as acetylcholine esterase inhibitors (e.g., tacrine, donepezil, galantamine, rivastigmin) and memantine;
13. Known history of allergies to tomatoes or tomato-based products;
14. High habitual intake of tomatoes, grapes, and tomato-based products confirmed by food frequency questionnaire (>5 times per day). Subjects who have high intake of these products are asked to take off these products for 4 weeks and after this washout period they will be reconsidered to participate in the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Evidence of improvement in memory after treatment with Fruitflow-II, resVida (Resveratrol), alone or in combination | 3 months
  The following tests will be used for evaluating cognitive function:
  1. Cambridge Neuropsychological Test Automated Battery (CANTAB). We use 5 tests which are mostly related to memory functioning including following:
     * Visual memory tests incuding (A) Paired Associates Learning (PAL) and (B) Pattern Recognition Memory (PRM)
     * Executive function, working memory and planning tests including (A) Stockings of Cambridge (SOC) and (B) Spatial Working Memory (SWM)
     * Semantic/verbal memory tests including (A) Verbal Recognition Memory (VRM)
  2. Trail-Making Test (TMT)
  3. Verbal Fluency Test

SECONDARY OUTCOMES:
Maximal VO2 (VO2 max) | 3 months
  Aerobic fitness (VO2 max) will be assessed by graded maximal exercise testing on a stationary bicycle. Oxygen uptake (VO2) will be measured from expired air samples to be taken at 30-s intervals until a maximal VO2 (VO2 max) is attained or to the point of test termination secondary to symptom limitation and/or volitional exhaustion. VO2 max will be defined as the highest recorded VO2 value when two of three criteria are satisfied: (1) a plateau in VO2 peak between two or more workloads; (2) a respiratory exchange ratio >1.00; and (3) a heart rate equivalent to their age-predicted maximum.
Blood Flow to the Brain | 3 months
  Cerebral blood flow velocity will be measured in the middle cerebral artery (MCA) and basilar artery (BA) using Transcranial Doppler ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Majid Fotuhi, MD, PhD, Principal Investigator — Memosyn Neurology Institute; Mehrnoosh Hadadi, MD, MPH, Study Director — Memosyn Neurology Institute
Locations (1):
- Memosyn Neurology Institute, 1205 York Road, Suite 11, Lutherville, Maryland, United States

REFERENCES:
- See also: Memosyn Neurology Institute — http://www.Memosyn.com